CLINICAL TRIAL: NCT00109486
Title: A Randomised, Double-Blind, Placebo-Controlled, Two-Week Crossover, Knemometric Assessment of the Effect of Fluticasone Furoate Nasal Spray 100mcg Once Daily on Short-Term Growth in Children Aged 6 to 11 Years With Seasonal and/or Perennial Allergic Rhinitis
Brief Title: Safety Study To Assess Growth In Children With Seasonal Allergic And/Or Perennial Allergic Rhinitis Treated With GW685698X Aqueous Nasal Spray Or Placebo Nasal Spray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FFR101747
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: GW685698X; seasonal allergic rhinitis; perennial allergic rhinitis; knemometry; children
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
The purpose of this study is to assess any effect in children with seasonal and/or perennial allergic rhinitis by GW685698X aqueous nasal spray (versus vehicle placebo nasal spray) on growth using knemometry.

ELIGIBILITY:
Inclusion criteria:

* Females (ages 6 to 11) who have not begun menses.
* Males (ages 6 to 12).
* Tanner Stage 1.
* History of SAR (Seasonal Allergic Rhinitis) or PAR (Perennial Allergic Rhinitis) of at least one year with either a current level of allergic rhinitis symptoms that warrants treatment and/or expected symptoms during a majority of the study period.
* Positive skin test to an appropriate seasonal or perennial allergen.

Exclusion criteria:

* History of abnormal growth or gross malnutrition.
* Clinically significant laboratory abnormality.
* History of any condition that may have substantially affected growth.
* Historical or current evidence of clinically significant, uncontrolled disease of any body system.
* Any asthma other than mild, intermittent asthma controlled by short-acting, beta-agonists.
* Recent major surgery and/or trauma to the legs.
* History of adrenal insufficiency.
* Current or prior treatment with any medication that may have a potential for an ongoing effect on linear growth.
* Use of corticosteroids, by any route, within 4 weeks prior to Visit 1.
* Any nasal condition or deformity that would impair nasal breathing or deposition of medication.
* Physical impairment that would affect the subject's ability to participate in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint will be the mean growth velocity (mm/wk) in lower leg growth, as determined by knemometry, over a 2-week treatment period with intranasal GW685698X aqueous nasal spray versus a 2-week treatment with placebo nasal spray.

SECONDARY OUTCOMES:
Secondary endpoints will include the frequency and type of clinical adverse events (AEs) experienced during treatment, nasal examinations, vital signs (systolic and diastolic blood pressure, heart rate [pulse]).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randers, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR101747 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register